CLINICAL TRIAL: NCT06438523
Title: A-prf,Nanochitosan Combined With A-prf Scaffold Compared to Chitosan in Vital Pulp Therapy for Symptomatic Irreversible Pulpitis of Mature Permanent Mandibular First Molar Teeth .Randomized Controlled Trials
Brief Title: A-prf,Nanochitosan Combined With A-prf Compared to Chitosan for Symptomatic Irreversible Pulpitis of Mature Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mai Sherif, Researcher, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29
Record Dates: First submitted 2024-05-15; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Pulpitis - Irreversible

STUDY DESIGN:
Intervention Model Description: Intervention:
  Intervention 1 : Vital pulp therapy using A-PRF as capping material. Intervention 2 : Vital pulp therapy using A-PRF mixed with Nano-Chitosan as capping material.
  Control/Comparator:
  Vital pulp therapy using Chitosan as capping material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Advanced Platelet rich fibrin,A-prf,A-PRF scaffold (Experimental): A-PRF will be prepared according to Choukroun's technique by drawing whole blood from the median cubital vein into a 10 ml plain plastic test tubes (non-citrated) without the addition of an anticoagulant reagent .
  To prevent the blood from coagulating, it will be centrifuged immediately using a table top centrifuge at 1500 rpm for 14 minute.
  Interventions: Procedure: PULPOTOMY OF MATURE PERMENANT TEETH
- A-prf mixed with nano chitosan (Experimental): A-PRF will be prepared according to Choukroun's technique by drawing whole blood from the median cubital vein into a 10 ml plain plastic test tubes (non-citrated) without the addition of an anticoagulant reagent .
  To prevent the blood from coagulating, it will be centrifuged immediately using a table top centrifuge at 1500 rpm for 14 minute then mixed with nanochitosan
  Interventions: Procedure: PULPOTOMY OF MATURE PERMENANT TEETH
- chitosan (Experimental): he access cavity will be prepared up to the level of pulp chamber floor using sterile round diamond bur size 1 in high-speed hand piece with coolant.Once the pulp has been reached, a sharp sterile excavator should be used to remove the pulp tissue to the level of the radicular/root canal orifices then chitosan will be applied
  Interventions: Procedure: PULPOTOMY OF MATURE PERMENANT TEETH

INTERVENTIONS:
Procedure: PULPOTOMY OF MATURE PERMENANT TEETH — Removal of coronal pulp and expose the orifices to apply the materials with aim to preserve vitality of remaining pulp

SUMMARY:
Clinical and radiographic assessment of A-prf,A-prf combined with nanochitosan compared to chitosan for symptomatic irreversible pulpits in lower permanent first molar

DETAILED DESCRIPTION:
3 groups are allocated using : Aprf Aprf combined with nanochitosan Chitosan

Each group will be subjected to tests:

Tooth sensibility via EPT (electrical pulp tester)and thermal test Radiolucency in digital radiograph Pain in NRS(6-12-24-72h)for 1 week

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Symptomatic irreversible pulpitis in mature mandibular molars only will be involved.

  * Patients of either gender aged from 15-30.
  * Tooth should give positive response to cold test.
  * Haemostasias should be achieved after total pulpotomy.
  * The tooth is restorable and free from advanced periodontal disease, cracks and splits.
  * Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
  * Patients who will agree to the consent and will commit to follow-up period.
  * Patients with mature root.
  * Patients with no internal or external resorption and no periapical lesions.
  * Soft tissues around the tooth are normal with no swelling or sinus tract.

Exclusion Criteria:

* Patients with immature roots.

  * Haemostasias after 10 minutes can not be controlled after total pulpotomy
  * Patients with any systemic disease that may affect normal healing.
  * Patients with periapical lesions or infections.
  * Pregnant females.
  * Patients who could/would not participate in a 6 months follow-up.
  * Patients with fistula or swelling
  * Patients with necrotic pulp.
  * Patients with old age.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-02 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
pain assessment | 6,12,24,72hours and 7 days postoperative
  Pain assessment using numerical rate scale

SECONDARY OUTCOMES:
Clinical and radiographic success | 1,3,6,9and 12 months
  It includes clinical and radiographic success if either of them failed the case will considered failed.
  Clinical failure :signs and symptoms of inflammation or infection Radiograph success and failure based on periapical index

CONTACTS AND LOCATIONS:
Overall Officials: wael H Kamel, Prof., Study Director — Future University in Egypt; Hani s sadek, Prof., Principal Investigator — Future University in Egypt
Locations (1):
- Future university, Cairo, Fifth Settlement, Egypt

IPD SHARING:
Plan to Share IPD: No